CLINICAL TRIAL: NCT02651883
Title: Effect of HPV Self-Collection on Cervical Cancer Screening in High Risk Women: My Body, My Test 3
Brief Title: Effect of Human Papillomavirus Self-Collection on Cervical Cancer Screening in High Risk Women: My Body, My Test 3
Acronym: MBMT-3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 14-3042; 1R01CA183891-01A1 (NIH)
Record Dates: First submitted 2016-01-04; First posted 2016-01-11 (Estimated); Last update posted 2022-12-02 (Actual); Status verified 2022-12

CONDITIONS: Cervical Cancer; Uterine Cervical Neoplasms; Human Papillomavirus
Keywords: Cervical cancer screening; HPV testing; Self-collection
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Self-Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Screening invitation (with education) (Active Comparator): Participants will receive a phone call providing (i) education on cervical cancer, and (ii) assistance scheduling an appointment for free cervical cancer screening at a study-affiliated clinic.
  Interventions: Behavioral: Screening invitation (with education)
- Self-collection for HPV testing (Experimental): Participants in the intervention arm will receive a kit to self-collect a sample and return it for HPV testing. Participants will then receive a phone call providing their HPV results plus (i) education on cervical cancer, and (ii) assistance scheduling an appointment for free cervical cancer screening at a study-affiliated clinic, if desired.
  Interventions: Behavioral: Screening invitation (with education); Behavioral: Self-collection for HPV testing

INTERVENTIONS:
Behavioral: Screening invitation (with education) — The participant will be provided with brief education about the importance and effectiveness of cervical cancer screening, and invited to schedule an appointment for a free in-clinic screening
  Other Names: Screening recall; Client reminder
Behavioral: Self-collection for HPV testing — Participant is provided with a kit to take a self-collected sample at home and return it by mail for HPV testing. Results are provided to participant by phone.
  Other Names: Self-testing; Self-sampling
  Arms: Self-collection for HPV testing

SUMMARY:
This study will investigate whether cervical cancer screening completion among under-screened women could be improved by offering HPV (human papillomavirus) testing by at-home self-collection followed by screening invitation compared to screening invitation alone.

DETAILED DESCRIPTION:
Invasive cervical cancer (ICC) is preventable through regular screening and treatment, but one fifth of US women report not receiving Pap testing at recommended intervals. More than half of ICC cases occur in these under-screened women. For women 30 years and older, the US Preventive Services Task Force recommends Pap smears alone every 3 years or physician-collected HPV testing with Pap smear (co-testing) every 5 years. The FDA approved primary HPV physician screening for US women 25 years and older. Self-collection for HPV testing is a valid and well-accepted method for detecting HPV infection with comparable sensitivity and specificity to physician-collection for detecting high-grade cervical lesions.

This 2-arm randomized control trial of 510 women will investigate whether offering HPV testing by mailed at-home self-collection to under-screened women increases their likelihood of completing cervical cancer screening. All participants will received a screening invitation by phone: a phone call providing (i) education on cervical cancer, and (ii) assistance scheduling an appointment for free screening at a study-affiliated clinic, if needed. Those randomized to the intervention arm will first be mailed a kit to self-collect a cervico-vaginal sample, return the sample for oncogenic HPV testing, and receive their results by phone. HPV negative women will be considered screening complete. HPV positive women will be invited to schedule an appointment for free follow-up in-clinic screening in the same call in which their results are delivered. The study endpoint of screening completion will be defined as completing in-clinic screening (control arm participants and HPV positive intervention arm participants) or receiving a negative HPV self-collection result (intervention arm).

Aim 1. Determine whether at-home HPV self-collection increases completion of cervical cancer screening among under-screened women offered enhanced reminders.

Aim 2. Examine possible mechanisms explaining the intervention's effect, or lack of an effect.

Aim 3. Estimate the incremental cost per additional woman completing screening of adding at-home HPV self-collection to enhanced reminders.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Aged 25 to 64 years old
* Living at ≤250% of the federal poverty line
* Eligible to receive cervical cancer screening from a study-associated clinic
* Resides within the same or bordering county of a study-associated clinic

Exclusion Criteria:

* Completion of cervical Pap screening in preceding 4 years
* Completion of HPV testing in preceding 6 years
* Pregnant
* History of hysterectomy
* Private insurance
* Unable to provide informed consent

Ages: 25 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 665 (Actual)
Dates: Start 2016-04; Primary Completion 2020-04-10 (Actual); Study Completion 2020-04-10 (Actual)

PRIMARY OUTCOMES:
Percent of participants that complete cervical cancer screening | Six months after enrollment
  Completion of cervical cancer screening is defined as (a) testing HPV negative by self-collection, or (b) completing in-clinic screening by i. HPV/Pap co-testing or ii. Pap smear alone.

SECONDARY OUTCOMES:
Levels of risk appraisal with regards to cervical cancer and screening | 1-5 weeks after completion of self-collection or screening invitation
  Risk appraisal will include multiple components measured by post-intervention questionnaire: Worry; Likelihood; Severity; Embodiment of risk (2 measures); "Gist" risk; Anticipated regret, action; Anticipated regret, inaction
Costs to payers | Throughout data collection period (average of 6 months per participant, approximately 3.5 years of study implementation)
  Incremental cost to payer (public or private) per additional woman screened
Level of intention to complete cervical cancer screening | 1-5 weeks after completion of self-collection or screening invitation
  As measured in post-intervention questionnaire
Level of self-efficacy to complete cervical cancer screening | 1-5 weeks after completion of self-collection or screening invitation
  As measured in post-intervention questionnaire
Percentage of participants who schedule a clinic appointment to get cervical cancer screening | 1-5 weeks after completion of self-collection or screening invitation
  Percent of participants that agree to schedule a clinic appointment to get a Pap smear or Pap/HPV co-testing

OTHER OUTCOMES:
Percentage of participants achieving primary outcome in different demographic categories | Throughout data collection period (average of 6 months per participant, approximately 3.5 years of study implementation)
  We will assess whether there are differences in the percentage of patients that complete cervical cancer screening by categories of age (e.g., younger than 45 vs. 45+), income, race, and educational level, measures collected at baseline
Prevalence of HPV mRNA (messenger ribonucleic acid) detection in self- and clinic-collected samples, abnormal cytology detected in clinic samples, and high-grade lesions (CIN2+) as detected in follow-up colposcopy screening (as indicated) | Throughout data collection period (average of 6 months per participant, approximately 3.5 years of study implementation)
  Prevalence of HPV infection (as determined by presence of hrHPV mRNA in self- and clinic samples), abnormal cytology (ASCUS+ per NCI Bethesda system), and high-grade lesions (CIN2+, as determined by follow-up colposcopic inspection with biopsy as indicated) will be determined from medical records (as permitted by HIPAA authorization) and compared between the arms
Percentage of patients referred to and completing colposcopy | Throughout data collection period (average of 6 months per participant, approximately 3.5 years of study implementation)
  Referral to and completion of colposcopy will be determined from medical records (as permitted by HIPAA authorization) and compared between the arms
Number of patients referred to and completing colposcopy | Throughout data collection period (average of 6 months per participant, approximately 3.5 years of study implementation)
  Referral to and completion of colposcopy will be determined from medical records (as permitted by HIPAA authorization) and compared between the arms
Number of patients referred to and completing treatment | Throughout data collection period (average of 6 months per participant, approximately 3.5 years of study implementation)
  Referral to and completion of treatment will be determined from medical records (as permitted by HIPAA authorization) and compared between the arms
Percentage of patients referred to and completing treatment | Throughout data collection period (average of 6 months per participant, approximately 3.5 years of study implementation)
  Referral to and completion of treatment will be determined from medical records (as permitted by HIPAA authorization) and compared between the arms
Attitudes towards HPV, cervical cancer, and cervical cancer screening | 1-5 weeks after completion of self-collection or screening invitation
  Attitudes will include multiple components measured by post-intervention questionnaire, including perceived barriers to screening, perceived benefits to screening, defensive processing of risk information, and subjective norms about screening

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer S Smith, PhD, Principal Investigator — UNC Chapel Hill
Locations (1):
- University of North Carolina Gillings School of Public Health, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ganguly AP, Pretsch PK, Brewer NT, Spees LP, Hudgens MG, Sanusi B, Barclay L, Carter A, Wheeler SB, Smith JS. Streamlined Self-Collection Screening for Sexually Transmitted Infections and Human Papillomavirus: A Single-Group Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2026 Jan 2;9(1):e2551345. doi: 10.1001/jamanetworkopen.2025.51345. PMID 41505134
- [Derived] Broshkevitch CJ, Pretsch PK, Spees LP, Wheeler SB, Sanusi B, Des Marais A, Barclay L, Carter A, Hudgens MG, Brewer NT, Smith JS. Underscreened Women's Reactions to At-Home Self-Collected Human Papillomavirus Test Result Delivery. Sex Transm Dis. 2026 Feb 1;53(2):109-115. doi: 10.1097/OLQ.0000000000002256. Epub 2025 Oct 21. PMID 41118505
- [Derived] Bukowski A, Smith JS, Wheeler SB, Sanusi B, McGuire FH, Zeno E, Des Marais AC, Barclay L, Hudgens MG, Jackson S, Brewer NT. Cervical Cancer Screening Knowledge, Perceptions, and Behaviors in a Multiracial Cohort of Low-Income, Underscreened Women in North Carolina. J Womens Health (Larchmt). 2023 Sep;32(9):970-981. doi: 10.1089/jwh.2022.0412. Epub 2023 Jun 16. PMID 37327372
- [Derived] Pretsch PK, Spees LP, Brewer NT, Hudgens MG, Sanusi B, Rohner E, Miller E, Jackson SL, Barclay L, Carter A, Wheeler SB, Smith JS. Effect of HPV self-collection kits on cervical cancer screening uptake among under-screened women from low-income US backgrounds (MBMT-3): a phase 3, open-label, randomised controlled trial. Lancet Public Health. 2023 Jun;8(6):e411-e421. doi: 10.1016/S2468-2667(23)00076-2. Epub 2023 May 11. PMID 37182529
- [Derived] Biddell CB, Spees LP, Smith JS, Brewer NT, Des Marais AC, Sanusi BO, Hudgens MG, Barclay L, Jackson S, Kent EE, Wheeler SB. Perceived Financial Barriers to Cervical Cancer Screening and Associated Cost Burden Among Low-Income, Under-Screened Women. J Womens Health (Larchmt). 2021 Sep;30(9):1243-1252. doi: 10.1089/jwh.2020.8807. Epub 2021 Apr 13. PMID 33851854
- [Derived] Spees LP, Des Marais AC, Wheeler SB, Hudgens MG, Doughty S, Brewer NT, Smith JS. Impact of human papillomavirus (HPV) self-collection on subsequent cervical cancer screening completion among under-screened US women: MyBodyMyTest-3 protocol for a randomized controlled trial. Trials. 2019 Dec 27;20(1):788. doi: 10.1186/s13063-019-3959-2. PMID 31881928